CLINICAL TRIAL: NCT00741884
Title: A Phase 2, Seven Week, Double-Blind, Placebo Controlled, Randomized, Parallel Group Study To Evaluate The Safety And Efficacy Of Three Doses Of A Controlled Release Formulation Of Varenicline For Smoking Cessation
Brief Title: A Study to Evaluate the Safety and Efficacy of Three Doses of a Controlled Release Formulation of Varenicline for Smoking Cessation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3051090
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 (Experimental)
  Interventions: Drug: Varenicline Controlled Release 1.2 mg
- Arm 2 (Experimental)
  Interventions: Drug: Varenicline Controlled Release 1.8 mg
- Arm 3 (Experimental)
  Interventions: Drug: Varenicline Controlled Release 2.4 mg
- Arm 4 (Active Comparator)
  Interventions: Drug: Varenicline Immediate Release 1 mg
- Arm 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline Controlled Release 1.2 mg — Varenicline CR tablet 1.2 mg BID for 7 weeks
  Arms: Arm 1
Drug: Varenicline Controlled Release 1.8 mg — Varenicline CR tablet 1.8 mg BID for 7 weeks
  Arms: Arm 2
Drug: Varenicline Controlled Release 2.4 mg — Varenicline CR tablet 2.4 mg BID for 7 weeks
  Arms: Arm 3
Drug: Varenicline Immediate Release 1 mg — Varenicline IR tablet 1 mg BID for 7 weeks
  Arms: Arm 4
Drug: Placebo — Placebo BID for 7 weeks
  Arms: Arm 5

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and tolerability of twice daily (BID) administration of three dose strengths (1.2 mg, 1.8 mg, and 2.4 mg) of varenicline controlled release (CR) tablets in adult smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cigarette smokers between the ages of 18 and 75 years, inclusive, who are motivated to stop smoking.
* Females of non-childbearing potential (surgically sterilized or at least 2 years postmenopausal) who are not nursing may be included.
* Subjects must have smoked an average of at least 10 cigarettes per day during the past year and over the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Subjects with clinically significant cardiovascular disease in the past 6 months.
* Subjects hospitalized within the past 12 months due to suicidal ideation or suicidal behavior or subjects considered to have serious suicidal ideation or suicidal behavior within the past 12 months.
* Subjects having active suicidal ideation or behavior identified at Screen or Baseline.
* Subjects currently or within the past 12 months requiring treatment for depression. Subjects with current or prior history of panic disorder, anxiety disorder, hostility or aggression disorder, perceptual/thinking disturbances, psychosis, or bipolar disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Continuous abstinence from smoking for weeks 4-7, carbon monoxide confirmed | 7 weeks

SECONDARY OUTCOMES:
7- day point prevalence of non-smoking at week 7 | 7 days
Scores on the Minnesota Nicotine Withdrawal Scale subscales | 7 weeks
Scores on the Modified Cigarette Evaluation Questionaire subscales | 7 weeks
PK analysis | 7 weeks
Safety Assessments: adverse events, C-SSRs, vital signs, body weight | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051090&StudyName=A%20study%20to%20evaluate%20the%20safety%20and%20efficacy%20of%20%20three%20doses%20of%20a%20controlled%20release%20formulation%20of%20varenicline%20for%20smoking%20cessation